CLINICAL TRIAL: NCT05257720
Title: Evaluation of the Role of Neurodegeneration in Treatment Resistant Schizophrenia With GFAP and S100B
Brief Title: Evaluation of the Role of Neurodegeneration in Schizophrenia
Status: Completed | Type: Observational
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Pelin Ozkara Menekseoglu, Medical Doctor, Istanbul Saglik Bilimleri University
Other Study IDs: 21-667
Record Dates: First submitted 2022-01-23; First posted 2022-02-25 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Schizophrenia
Keywords: schizophrenia, neurodegeneration, s100b, gfap
MeSH Terms: conditions — Schizophrenia; Nerve Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Remission: Patient with schizophrenia in remission
  Interventions: Diagnostic Test: GFAP, S100B
- treatment resistant: patient with treatment resistant schizophrenia
  Interventions: Diagnostic Test: GFAP, S100B
- controls: healthy controls
  Interventions: Diagnostic Test: GFAP, S100B

INTERVENTIONS:
Diagnostic Test: GFAP, S100B — It is planned to measure serum GFAP and S100 B protein levels by ELISA method.

SUMMARY:
Schizophrenia is a progressive psychiatric disorder with a lifetime prevalence of 1%, its etiology is not fully understood, and it progresses with relapses. There are significant differences between patients in the age of onset, frequency of attacks, response to treatment, and clinical course of the disease. Failure to respond adequately to treatment is defined as resistance to treatment and poses a great challenge in the clinical management of the disease, but the exact cause of treatment resistance has not been clarified yet. Neurodevelopmental hypothesis, neurodegenerative hypothesis, stress-diathesis hypothesis are some of them. In the neurodegenerative hypothesis, it is thought that biochemical changes cause chronic and progressive disorders of the nervous system, and schizophrenia is considered as one of these disorders. S100B, one of the biomarkers released from the central nervous system, is a glycoprotein synthesized by astrocytes; At low concentration, it ensures neuron survival, while at high concentration it causes neuronal cell apoptosis and is associated with neurodegeneration. GFAP on the other hand, can be measured in serum in proportion to the degree of damage by passing into the bloodstream as a result of astrocyte damage. It has been shown that these markers are associated with neurodegenerative diseases, autoimmune diseases and cerebrovascular pathologies and can be measured at a significant level in the blood. As far as is known, neurodegeneration has been found in patients with schizophrenia; however, there are not enough studies in the literature regarding the relationship of this neurodegeneration with treatment response and resistance. In recent years, many biomarker studies related to schizophrenia have been conducted. These studies continue in many different areas such as the early diagnosis of schizophrenia, the treatments to be applied after diagnosis, the response to the treatment given, and the clinical course of the disease, but no biomarker indicating the desired results has yet been found. In this study, measurement of s100B and GFAP serum levels in patients with treatment-resistant schizophrenia, remission schizophrenia and healthy controls, and evaluation of their relationship with response to treatment; Thus, it is aimed to investigate these points that have not been fully elucidated in the pathogenesis of schizophrenia and their use as biomarkers in predicting the response to treatment.

DETAILED DESCRIPTION:
Schizophrenia is a progressive and complex psychiatric disorder with a lifetime prevalence of 1%, usually diagnosed between the ages of 20-25, its etiology is not fully understood, and it progresses with relapses. In addition to positive symptoms such as delusions, hallucinations, disorganized speech and behavior, and negative symptoms such as affective blunting, anhedonia, and avulsion, impairment in social and occupational functionality and cognitive impairment can be observed.

The incidence of schizophrenia in relatives of individuals with schizophrenia is higher than in the general population. Although heredity is a strong component in the etiology of schizophrenia, environmental exposures and stressors such as maternal immune infection, obstetric complications, childhood trauma and cannabis exposure also play a role in the development and neuropathology of the disease. Hereditary risk and the interactions of these exposures with the genomic sequence form the basis of the neurodevelopmental hypothesis of schizophrenia.

The neurodevelopmental hypothesis proposes that disruption of brain development early in life is responsible for the onset of symptoms. According to the neurodevelopmental hypothesis, although the biological changes and other features of the disease are present in the patient long before the onset of the characteristic symptoms of schizophrenia, these symptoms will not appear in the patient until a certain level of development is reached by interacting with some factors.

Detection of some brain findings such as decreased cortical volume, ventricular enlargement, and altered gyrification patterns in the imaging findings in the initial period of schizophrenia supports the view that some changes in the brain can be seen even before the onset of schizophrenia, but in this view, no worsening of the damage in the brain is expected. Therefore, the neurodevelopmental model falls short of addressing the progressive brain damage observed in patients with chronic schizophrenia Studies show a worsening clinical course in 60% of patients with schizophrenia. The neurodegenerative hypothesis focuses on the fact that biochemical changes in schizophrenia are characterized by chronic and progressive impairment of the nervous system, leading to different clinical syndromes, loss of neurological function and behavioral disorders. It is thought that the presence of changes in the brain morphology of patients with schizophrenia in various studies indicates degeneration. In brain imaging, changes such as decrease in temporal lobe and frontal lobe volume, enlargement in the lateral ventricles and third ventricle, hippocampal atrophy have been detected. Changes in these areas of the brain indicate loss of white and gray matter. Detection of these differences in the first psychotic attacks and early-onset patients; suggests that the degenerative process starts from the earliest stages of the disorder. In addition, it has been shown that the difference between brain imaging of healthy controls and patients with schizophrenia increases with age.

Following the clinical onset of schizophrenia, patients differ significantly in disease course. Relapse is associated with significant psychological and social distress as well as increased economic burden in patients with schizophrenia and their families. Good response to antipsychotic drug and low optimal antipsychotic dose in patients with first episode schizophrenia; This suggests that relapse reduces drug response, and that the increase in the number of attacks is associated with resistance to treatment in schizophrenia. The state of not responding adequately to treatment is defined as resistance to treatment, and the most comprehensive definition of the concept of Treatment-Resistant Schizophrenia (TFS) was made by Kane, and it was named "Kane Criteria". Kane Criteria Criteria for resistance to treatment applied in the past; Failure to respond to at least three antipsychotic treatments at 1000mg/day chlorpromazine or equivalent dose for six weeks in the previous five years. Lack of a good functioning period in the last five years. Criterion of severity of psychopathology; A Brief Psychiatric Rating Scale (BPRS) score of 45 and above, At least two of the 4 positive symptoms of BPRS (thought disorientation, skepticism, hallucinatory behavior, unusual thoughts) are 4 and above, Clinical General Impression (CGI) score is 4 and above Prospective treatment non-response criteria; Unresponsive to haloperidol therapy up to 60 mg/day. (Response to treatment was defined as a BPRS score of more than 20% and a CGI score of 3 or less, or a BPRS score of 35 or less). Diagnosis of Treatment-Resistant Schizophrenia in Clinical Practice - A history of two antipsychotic treatments - At least 6 weeks on an antipsychotic and at least 600 mg Chlorpromazine equivalent dose - Brief Psychiatric Rating Scale (CPRS) ≥45 - Positive and Negative Syndrome Global Scale (PANNS) ≥75 - Clinical Impression Scale-Severity of Disease (CGI-HȘ) ≥ 4 - General Evaluation of Functioning (IGD) ≤50 In psychiatry, the diagnosis is made based on the evaluation of signs and symptoms in the clinical interview, and there is no biological "gold standard" diagnosis. It has been shown that in patients with first episode schizophrenia, each episode lasts longer than the previous episode, and relapse is associated with progressive loss of cortical tissue and brain volume. Relapse is an expression of worsening psychopathology and it is thought that some neurobiological pathways may cause relapse. The glial fibrillary acidic protein GFAP, which is one of the reactive astrocyte-specific biomarkers indicating astrogliosis, is not released from the healthy astrocyte. The increase in GFAP indicates damage and inflammation in the astrocyte. It is also secreted in different amounts from different parts of the brain. GFAP can be measured in serum in proportion to the degree of damage by passing into the blood circulation as a result of astrocyte damage. One of the cytoskeletal components (GFAP), it has been associated with neurodegenerative diseases such as Alzheimer's and amyotrophic lateral sclerosis, and is thought to play a role in the etiology of schizophrenia and is one of the potential markers of neurodegeneration and progression in schizophrenia. In a study measuring the amount of serum GFAP in patients with schizophrenia and healthy volunteers, GFAP was found to be high in the schizophrenia group, but it was noted that it was higher especially in patients using clozapine.

The S100B protein is a member of the calcium-binding protein group and is secreted from many cells, such as astrocytes, oligodendrocytes, certain neuronal populations, adipocytes, or lymphocyte populations. This protein is released from stimulated or damaged astrocytes into the cerebrospinal fluid (CSF) and crosses the blood-brain barrier and enters the peripheral circulation. The S100B protein (depending on its level) can have a trophic or toxic effect on surrounding neurons, astrocytes, or microglia. At low concentration, S100B ensures neuron survival, but at higher level it leads to neuronal cell apoptosis and is associated with brain damage or neurodegeneration. Various brain tumors, neuroinflammatory and neurodegenerative disorders, psychiatric diseases and even major cardiac events have been investigated. Serum and cerebrospinal concentrations of S100B are found to be high in schizophrenia, which is thought to indicate activation of astrocytes or loss of oligodenrocytes. Studies in cell culture and experiments with ligands have shown that S100B can increase dopaminergic neurotransmission. With the pathogenesis of the disease, varying concentrations of S100B in patients with schizophrenia; It is thought that the binding of S100B to the D2 receptor leads to a decrease in glutamate concentration at synapses as a result of increased signal transduction and increased glutamate uptake in astrocytes, and may also be related to the role of S100B in neuronal apoptosis in many different ways.

Data Collection and Evaluation Scales

1. Sociodemographic and Clinical Data Form:
2. The Brief Psychiatric Rating Scale (BPRS)
3. Positive and Negative Syndrome Scale (PANSS)
4. Clinical Global Impression (CGI)
5. General Evaluation of Functioning (IGD)
6. STANDARDIZED MINI MENTAL TEST (SMMT) or MODIFIED MINI MENTAL TEST (MMSE-E) FOR THE UNEDUCTED

ELIGIBILITY:
Inclusion Criteria for Patients

* Being between the ages of 18-65
* Being at least primary school graduate
* Not having mental retardation
* Not having visual and hearing problems that affect communication
* Having a diagnosis of schizophrenia according to DSM-5 criteria
* Absence of comorbid psychiatric disease
* Systemic and/or systemic disease. or neurological (such as hypertension, diabetes mellitus, infection, dementia, epilepsy, Parkinson's disease, cardiovascular, renal, urological, hepatic, pulmonary, genetic, endocrine diseases, nutritional disorders, intoxications, operations, and other organic disorders), S100B and GFAP levels No medical condition known to affect it
* No history of head trauma
* No alcohol and/or substance use disorder
* Body mass index (BMI) > 18 kg/m2 , BMI < 25 kg/m2
* Not having been diagnosed with metabolic syndrome
* 1. and/or No 2nd degree relatives with schizophrenia and/or a similar psychiatric disorder
* After being informed about the study,

Inclusion Criteria for Healthy Controls

* Being between the ages of 18-65
* Being at least primary school graduate
* Not having mental retardation
* Not having vision and hearing problems that affect communication
* Among first and/or second degree relatives No history of schizophrenia and/or any other psychiatric disease
* Systemic and/or neurological (hypertension, diabetes mellitus, infection, dementia, epilepsy, parkinson's disease, cardiovascular, renal, urological, hepatic, pulmonary, genetic, endocrine diseases, nutritional disorders, intoxications , operations and other organic disorders), absence of medical conditions known to adversely affect S1000B and GFAP levels
* No history of head trauma
* No alcohol and/or substance use disorder
* Body mass index (BMI)> 18 kg/m2 , < 25 kg/ m2
* Not having been diagnosed with metabolic syndrome
* Having a 1st and/or 2nd degree relatives with schizophrenia and/or similar No psychiatric disorder
* Having consented to participate in the study after being informed about the study Exclusion Criteria
* Not between the ages of 18-65
* Having a diagnosis of mental retardation
* Having vision and/or hearing problems that affect communication
* Presence of psychiatric illness
* First and/or second degree relatives between schizophrenia and/or another psychiatric disease diagnosis
* Systemic and/or neurological (hypertension, diabetes mellitus, infection, dementia, epilepsy, parkinson's disease, cardiovascular, renal, urological, hepatic, pulmonary, genetic, endocrine diseases, nutritional disorders, intoxications, operations and other organic disorders), presence of medical conditions known to adversely affect S100B and GFAP levels
* Presence of non-psychiatric drug use
* Presence of head trauma
* Presence of alcohol and/or substance use disorder
* Body mass index (BMI) > 25 kg /m2
* Metabolic syndrome being diagnosed as Having schizophrenia and/or a similar psychiatric disorder in 1st and/or 2nd degree relatives
* After being informed about the study, the patient and/or his guardian or healthy control did not give consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Our research was planned to recruit 60 patients with schizophrenia in remission, 60 patients with treatment-resistant schizophrenia, and 60 healthy volunteers, followed by Mazhar Osman Bakırköy Psychiatry Training and Research Hospital TRSMs and/or inpatient units, according to the inclusion and exclusion criteria. Consent will be obtained from all patients and healthy volunteers participating in the study with an informed consent form that provides information about the purpose of the study.
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
serum GFAP levels | 6 months
  It is planned to measure serum GFAP levels by ELISA method.
serum S100 B protein levels | 6 months
  It is planned to measure serum S100 B protein levels by ELISA method.

CONTACTS AND LOCATIONS:
Locations (1):
- T.C. Sağlik Bilimleri Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker E, Kestler L, Bollini A, Hochman KM. Schizophrenia: etiology and course. Annu Rev Psychol. 2004;55:401-30. doi: 10.1146/annurev.psych.55.090902.141950. PMID 14744221
- [Background] Khavari B, Cairns MJ. Epigenomic Dysregulation in Schizophrenia: In Search of Disease Etiology and Biomarkers. Cells. 2020 Aug 5;9(8):1837. doi: 10.3390/cells9081837. PMID 32764320
- [Background] Buoli M, Serati M, Caldiroli A, Cremaschi L, Altamura AC. Neurodevelopmental Versus Neurodegenerative Model of Schizophrenia and Bipolar Disorder: Comparison with Physiological Brain Development and Aging. Psychiatr Danub. 2017 Mar;29(1):24-27. doi: 10.24869/psyd.2017.24. PMID 28291970
- [Background] Pino O, Guilera G, Gomez-Benito J, Najas-Garcia A, Rufian S, Rojo E. Neurodevelopment or neurodegeneration: review of theories of schizophrenia. Actas Esp Psiquiatr. 2014 Jul-Aug;42(4):185-95. Epub 2014 Jul 1. PMID 25017496
- [Background] Kochunov P, Hong LE. Neurodevelopmental and neurodegenerative models of schizophrenia: white matter at the center stage. Schizophr Bull. 2014 Jul;40(4):721-8. doi: 10.1093/schbul/sbu070. Epub 2014 May 27. PMID 24870447
- [Background] Schnieder TP, Dwork AJ. Searching for neuropathology: gliosis in schizophrenia. Biol Psychiatry. 2011 Jan 15;69(2):134-9. doi: 10.1016/j.biopsych.2010.08.027. Epub 2010 Oct 30. PMID 21035789
- [Background] Takeuchi H, Siu C, Remington G, Fervaha G, Zipursky RB, Foussias G, Agid O. Does relapse contribute to treatment resistance? Antipsychotic response in first- vs. second-episode schizophrenia. Neuropsychopharmacology. 2019 May;44(6):1036-1042. doi: 10.1038/s41386-018-0278-3. Epub 2018 Nov 22. PMID 30514883
- [Background] Cooper JD, Han SYS, Tomasik J, Ozcan S, Rustogi N, van Beveren NJM, Leweke FM, Bahn S. Multimodel inference for biomarker development: an application to schizophrenia. Transl Psychiatry. 2019 Feb 11;9(1):83. doi: 10.1038/s41398-019-0419-4. PMID 30745560
- [Background] Pillai A, Schooler NR, Peter D, Looney SW, Goff DC, Kopelowicz A, Lauriello J, Manschreck T, Mendelowitz A, Miller DD, Severe JB, Wilson DR, Ames D, Bustillo J, Kane JM, Buckley PF. Predicting relapse in schizophrenia: Is BDNF a plausible biological marker? Schizophr Res. 2018 Mar;193:263-268. doi: 10.1016/j.schres.2017.06.059. Epub 2017 Jul 19. PMID 28734907
- [Background] Kim R, Healey KL, Sepulveda-Orengo MT, Reissner KJ. Astroglial correlates of neuropsychiatric disease: From astrocytopathy to astrogliosis. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Dec 20;87(Pt A):126-146. doi: 10.1016/j.pnpbp.2017.10.002. Epub 2017 Oct 6. PMID 28989099
- [Background] Rodrigues-Amorim D, Rivera-Baltanas T, Del Carmen Vallejo-Curto M, Rodriguez-Jamardo C, de Las Heras E, Barreiro-Villar C, Blanco-Formoso M, Fernandez-Palleiro P, Alvarez-Ariza M, Lopez M, Garcia-Caballero A, Olivares JM, Spuch C. Plasma beta-III tubulin, neurofilament light chain and glial fibrillary acidic protein are associated with neurodegeneration and progression in schizophrenia. Sci Rep. 2020 Aug 31;10(1):14271. doi: 10.1038/s41598-020-71060-4. PMID 32868793